CLINICAL TRIAL: NCT07326696
Title: Thoracic Thrust With Cervical Non-Thrust Mobilization in Mechanical Neck Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FUI/CTR/2025/23
Record Dates: First submitted 2025-12-26; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Chronic Mechanical Neck Pain
Keywords: neck pain; chronic neck pain; mechanical neck pain
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participant will be blinded to the allocation of treatement groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A; thoracic thrust (Experimental): thoracic thrust in addition to standard treatment
  Interventions: Procedure: Group A:Thoracic thrust
- Group B: cervical non-thrust mobilization (Active Comparator): standard treatment of cervical non-thrust mobilization and home-based therapeutic exercises
  Interventions: Procedure: Group B: Cervical non thrust mobilization

INTERVENTIONS:
Procedure: Group A:Thoracic thrust — Group A will receive manipulation protocol as addition to standard treatment. Manipulation protocol:
  High velocity, low amplitude as described by Maitland on thoracic hypomobile segments (T1-6)
  Therapeutic exercise protocol:
  Cervical and thoracic mobility exercises.
  Arms: Group A; thoracic thrust
Procedure: Group B: Cervical non thrust mobilization — Intervention:
  Group B will receive mobilization, post-facilitation stretch and exercise protocol.
  Mobilization protocol:
  Grade III or IV mobilization as described by Maitland on cervical Hypomobile segments (C2-7)
  Therapeutic exercise protocol:
  Cervical and thoracic mobility exercises.
  Arms: Group B: cervical non-thrust mobilization

SUMMARY:
This study is a randomised controlled trial and the purpose of this study is to determine the effects of thoracic thrust with cervical non-thrust mobilization in mechanical neck pain on components such as pain, thoracic range of motion, kyphotic angle, craniovertebral angle and proprioception.

DETAILED DESCRIPTION:
Particiapants will be divided into two groups through coin toss method, one group will recieve thoracic manipulation as addition to cervical mobilization and therapeutic exercises.

ELIGIBILITY:
Inclusion criteria:

* Both male and female
* Age: 20-40 years
* Numeric pain rating scale (3<) (13)
* Neck pain for more than 3 months
* Cervical hypomobility (C2-C7)
* Thoracic hypomobility (T1-T6)
* CranioVertebral Angle < 48 Degrees

Exclusion criteria:

* Serious pathology (e.g. neoplasm, fracture)
* History of whiplash injury within the past 6 months
* Cervical spinal stenosis
* Radiculopathy
* Neurological deficit
* Structural deformities
* Vertebrobasilar artery insufficiency
* Pregnancy
* Prior surgery of cervical or thoracic spine

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 46 (Estimated)
Dates: Start 2025-01-25 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-01-15 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity | baseline, 1st and 2nd week
  Pain will be assessed by Numeric pain scale rating (NPRS).It is numeric 11-point scale, with 0 meaning no pain and 10 being worst pain.
Thoracic kyphosis | baseline, 1st week and 2nd week
  Thoracic Kyphosis is measured by Inclinometer. It is measured via summation of angles of two inclinometers, placed on anatomical landmarks (T1-3-12).
Thoracic Range of Motion | baseline, 1st week, 2nd week
  Thoracic ROM (rotation) is measured by Inclinometer. Measured by placing the inclinometer at T1 segment with participant in a lumbar locked position.
Craniovertebral angle | baseline,1st week, 2nd week
  Craniovertebral angle (CVA)is measured by Goniometer. it is Angle measured between tragus of ear and C7 spinous process.
Proprioception | baseline, 1st and 2nd week
  Proprioception is measured by Joint position sense/ error test. Participant wears a laser mounted headband and performs active neck movements with eyes closed on a target.

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation University College of Physical Therapy, Islamabad, Punjab Province, Pakistan